CLINICAL TRIAL: NCT06341543
Title: Use of QuantiFERON® CMV in the Therapeutic Decision in Asymptomatic CMV Infection in Solid Organ Transplant Recipients
Brief Title: Quantiferon CMV to Identify Treatment Need for Asymptomatic CMV Infection After Solid Organ Transplant (QUANTIFOT)
Acronym: QUANTIFOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QUANTIFOT; PHRCI-2021-68 (Other Grant/Funding Number: DGOS (France))
Record Dates: First submitted 2024-03-18; First posted 2024-04-02 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cytomegalovirus Infections; Heart Transplantation; Kidney Transplantation; Lung Transplantation; Liver Transplantation
Keywords: solid organ transplantation; cytomegalovirus; CMV; quantiferon; IGRA; interferon gamma release assay; antiviral; adverse effect; viremia
MeSH Terms: conditions — Cytomegalovirus Infections; Viremia | interventions — Fees and Charges

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qantiferon CMV result communicated to the clinician in charge (Experimental): In this arm, the result of the CMV-QF will be communicated to the clinician in charge. If QF-CMV is positive, the clinician will be advised not to treat the patient. If QF-CMV is negative, he/she will be advised to use or not antiviral therapy, according to the guidelines and the local practice.
  Interventions: Diagnostic Test: Quantiferon CMV (assay that determine the presence of CMV-specific T lymphocytes).; Other: Communication of the result of the QF-CMV to the clinician in charge
- Qantiferon CMV result NOT communicated to the clinician in charge (Other): In this arm, the result of the CMV-QF will NOT be communicated to the clinician in charge. He/she will be advised to use or not antiviral therapy, according to the guidelines and the local practice.
  Interventions: Diagnostic Test: Quantiferon CMV (assay that determine the presence of CMV-specific T lymphocytes).

INTERVENTIONS:
Diagnostic Test: Quantiferon CMV (assay that determine the presence of CMV-specific T lymphocytes). — The QF-CMV will be performed in all participants.
Other: Communication of the result of the QF-CMV to the clinician in charge — The result of the CMV-QF will be communicated to the clinician in charge only for the patients randomised in the group "communication of the QF-CMV result to the clinician in charge".
  Arms: Qantiferon CMV result communicated to the clinician in charge

SUMMARY:
Context

Cytomegalovirus (CMV) infection is a frequent and potentially severe event in solid organ transplant (SOT) recipients.

Most of available treatment display adverse effects that limit their use. Therefore, in case of an infection, it is of primary importance to identify the patients at high risk of severe infection and/or disease, and who ill benefit the most from antiviral therapy.

As CMV infection is mainly controlled by cellular immunity, measuring specific anti-CMV T lymphocyte immunity could be an interesting tool for identifying these at-risk individuals. One of these tests is the QuantiFERON-CMV (QF-CMV) assay (QuiagenTM, Courtabœuf, France).

Aim of the study

The aim of the study is to determine the extent to which the QF-CMV can be use to identify, among SOT recipients with a CMV viremia, those that may not need antiviral therapy.

Methods

Participation to the study will be proposed to SOT recipients with an asymptomatic CMV infection with a blood viral load between 1,000 and 15,000 IU/mL.

The QF-CMV will be performed in included participants, and the result will be given or not to the clinician in charge (according to the attributed group through randomisation).

* In the group without result communication, the clinician in charge will determine whether a treatment is needed according to the guidelines and the local practices.
* in the group with result communication, the clinician in charge will be advised not to introduce antiviral therapy if the result is positive, and to determine whether a treatment is needed according to the guidelines and the local practices if the result is positive.

In the following weeks, the viral load will be monitored, along with creatininemia, cell blood count, and kalemia (to detect antiviral adverse effect).

The participants will be sampled:

* 5 to 12 days after QF-CMV sampling (V2) ;
* 7 to 14 days days after V2 (V3 - between D12 and D26) ;
* 7 to 14 days days after V3 (V4 - between D19 and D40) .

Endpoints

The primary endpoint is the rate of uncontrolled infection 5 to 12 days after QF-CMV sampling, defined as follows:

* Blood CMV viral load >10,000 IU/mL [4 log];
* And/or increase in blood viral load ≥0.5 log IU/mL with CV otherwise >5000 IU/mL;
* And/or the onset of CMV disease.

The secondary endpoint is the is the occurrence antiviral adverse effects (hematoxicity or nephrotoxicity).

DETAILED DESCRIPTION:
Context.

Solid organ transplant (SOT) recipients are at high risk of opportunistic infections, particularly due to cytomegalovirus (CMV).

Regarding CMV infection after transplantation, two approaches are possible: either antiviral prophylaxis for several months, followed by monitoring of blood CMV viral load (or viremia), or immediate monitoring of viral load without prophylaxis.

In both cases, the detection of a CMV viral load raises a complex question: is antiviral treatment necessary? Indeed, not all viremia leads to CMV disease: some patients spontaneously control their viremia.

In order to limit unnecessary treatments, their toxicity and their cost, new tools are needed to identify people at high risk of developing a high viral load or CMV disease.

As CMV infection is mainly controlled by cellular immunity, measuring specific anti-CMV T lymphocyte immunity could be an interesting tool for identifying these at-risk individuals.

The QuantiFERON-CMV (QF-CMV) test (QuiagenTM, Courtabœuf, France) is an interferon-gamma (IFN-γ) release assay (IGRA), which measures the presence of anti-CMV T lymphocyte immunity. Results from previous retrospective studies suggest that in cases of CMV replication, it may be relevant to base the therapeutic attitude not only on the virological characteristics of this replication, but also on the existence of specific T lymphocyte immunity.

The aim of this study is therefore to prospectively assess the contribution of QF-CMV to therapeutic decisions in cases of intermediate CMV viral load (between 1,000 and 15,000 IU/mL).

Methods

SOT recipients with a detectable blood CMV viral load (CV1) between 1,000 and 15,000 IU/mL without symptoms (fever, organ damage) will be offered participation in the study within 48 hours of detection of this CMV viral load.

After inclusion, participants will be immediately sampled for QF-CMV.

They will be randomized (2:1) into 2 groups:

* An experimental group in which the result of the QF-CMV will be communicated to the doctor in charge;
* A control group in which the result is not reported to the doctor in charge.

In the experimental group, the recommended attitude will depend on the QF-CMV result:

* If positive, the physician in charge will be advised not to introduce antiviral treatment;
* If is negative or indeterminate, the physician in charge will be advised to proceed according to the standard of care. He/she will be free to introduce or not the antiviral molecule of his choice.

In the control group, the physician in charge will be advised to proceed according to the standard of care, based on current recommendations and local practices.

In both groups, as routinely done when a CMV viral load is detected in the blood, this parameter will be checked several times after the 1st detection (V0):

* 5 to 12 days after QF-CMV sampling (CV - V2 = D5 to D12) ;
* 7 to 14 days after CV2 (CV3 - V3 = D12 to D26) ;
* 7 to 14 days after CV3 (CV4 - V4 = D19 to D40). Similarly, blood cell count, kalemia and creatininemia were performed at baseline and then at V2, V3 and V4.

The primary endpoint is the rate of uncontrolled infection at 5 to 12 days after QF-CMV sampling (V2), defined as follows:

* Blood CMV viral load >10,000 IU/mL [4 log] ;
* And/or increase in blood viral load ≥0.5 log IU/mL with CV otherwise >5000 IU/mL ;
* And/or the onset of CMV disease.

Conversely, the blood CMV viral load will be considered controlled if its value at V2 does not exceed 10,000 IU/mL [4 log] and :

* It decreases (regardless of the magnitude of the decrease);
* Or increases, but by less than 0.5 log IU/mL ;
* or is stable. In the event of uncontrolled infection at V2, the physician in charge should manage the viral load in accordance with current recommendations and local practices (in most cases, antiviral treatment should be introduced if this has not already been done), and continue monitoring at V3 and V4. He will be free to introduce or not the antiviral molecule of his choice.

In the event of controlled infection at V2, the physician in charge will be advised not to initiate antiviral treatment if this has not already been done, and to continue monitoring at V3 and V4.

The secondary endpoint is the occurrence of an iatrogenic event (hematoxicity or nephrotoxicity) related to antivirals; parameters that may reflect such toxicity (blood cell count, kalemia, creatinin) will be collected at inclusion (V1) and then at the 3 times mentioned above (V2 to V4).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Solid organ transplant recipient (heart, kidney, liver and lung)
* Detectable CMV viral load between 1,000 and 15,000 IU/mL (including 2 borderline values):

  * Asymptomatic (no fever or organ dysfunction) ;
  * Occurrence within 2 years of transplantation in the absence of primary post-transplant anti-CMV prophylaxis;
  * Or within 2 years of discontinuation of primary post-transplant anti-CMV prophylaxis if such prophylaxis was used.
* Having signed an informed consent form.
* Affiliated to a social security scheme.

Exclusion Criteria:

* Presence of anti-Herpesviridae treatment when CMV replication is detected ([val]aciclovir, [val]ganciclovir, foscarnet, cidofovir, letermovir, maribavir, anti-CMV immunoglobulins, cidofovir, brincidofovir).
* Pregnant or breast-feeding women.
* Persons under guardianship or trusteeship.
* Subjects under administrative or judicial supervision.
* Subject unable to be contacted in case of emergency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
proportion of participants with CMV viral load (>10,000 IU/mL, or increase ≥0.5 log IU/mL) | 5 to 12 days after QF-CMV sampling, and up to 40 days after first CMV detection
  Uncontrolled infection 5 to 12 days after QF-CMV sampling is defined as follows:
  * Blood CMV viral load >10,000 IU/mL [4 log];
  * And/or increase in blood viral load ≥0.5 log IU/mL with CV otherwise >5000 IU/mL
proportion of participants with CMV disease | 5 to 12 days after QF-CMV sampling, and up to 40 days after first CMV detection
  CMV disease is defined as follows:
  * pneumonia onset
  * colitis onset
  * encephalitis onset
  * hepatitis onset

SECONDARY OUTCOMES:
proportion of participants with antiviral-associated anemia | 5 to 12 days after QF-CMV sampling, and up to 40 days after first CMV detection
  hemoglobin <110 g/L or decrease >10%
proportion of participants with antiviral-associated leucopenia | 5 to 12 days after QF-CMV sampling, and up to 40 days after first CMV detection
  PNN <1000/mm3 or decrease >30%
proportion of participants with antiviral-associated thrombopenia | 5 to 12 days after QF-CMV sampling, and up to 40 days after first CMV detection
  platelets <130 G/L or decrease >20%
proportion of participants with antiviral-associated tubulotoxicity (hypokaliemia) | 5 to 12 days after QF-CMV sampling, and up to 40 days after first CMV detection
  kaliemia <3,5 mMol
antiviral-associated kidney failure (creatininemia) | 5 to 12 days after QF-CMV sampling, and up to 40 days after first CMV detection
  creatininemia increase >20%

CONTACTS AND LOCATIONS:
Overall Officials: Martine Pernollet, Study Chair — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Grenoble, Maryland, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification, will be available beginning 3 months and ending 5 years following article publication.
  Researchers who provide a methodologically sound proposal.will be given access to these data. data requestors will need to sign a data access agreement.
  Proposals should be directed to oepaulard@chu-grenoble.fr
Supporting Information: CSR
Time Frame: beginning 3 months and ending 5 years following article publication.
Access Criteria: beginning 3 months and ending 5 years following article publication.
  Researchers who provide a methodologically sound proposal.will be given access to these data.